CLINICAL TRIAL: NCT01492621
Title: White Matter Structure and Response to Treatment With Antidepressants: a Study of Desvenlafaxine in Major Depression. A Pilot Study
Brief Title: Effect of Antidepressants on White Matter Structure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Valerie Tourjman, Associate director of clinical research, Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DTI
Record Dates: First submitted 2011-12-12; First posted 2011-12-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Major Depression
Keywords: major depression; DTI; inflammatory markers; cognition
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Desvenlafaxine — Desvenlafaxine 50mg from week 1-8. At week 8 optional increase to 100mg if remission has not been attained.
  Other Names: Pristiq

SUMMARY:
Subjects with major depression will be evaluated and intensively characterized through questionnaires, computerized cognitive evaluation and laboratory investigations. Magnetic resonance imaging will be used to document baseline white matter structure. subjects will then receive desvenlafaxine which will be adjusted as clinically indicated. After 16 weeks the evaluations will be repeated.

DETAILED DESCRIPTION:
40 subjects will be included in the study. Diagnosis will be confirmed by MINI. Participants will be characterised using questionnaires, pain threshold, cognition, facial expression recording and MRI. Desvenlafaxine will be initiated at 50mg AM. At week 8 Desvenlafaxine may be increased to 100mg as clinically indicated. Measures will be repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Major depression
* Age 18 to 55
* Hamilton grater or equal to 20

Exclusion Criteria:

* Major neurologic disorder
* Major cardiovascular disorder
* Unstable medical condition
* Significant psychiatric co-morbidity
* Current substance dependance
* Pregnancy or lactation -Treatment resistance as defined by nonresponse to 2 or more antidepressant treatments (adequate dose and duration) -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-09 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Anisotropy | 16 weeks
  Degree of anisotropy will be measured at baseline and 16 weeks and correlated to remission status

SECONDARY OUTCOMES:
cognitive measures | 16 weeks
  cognitive deficits will be measured at baseline and 16 weeks and correlated to anisotropy using computerized neuropsychological testing of memory, speed and executive function.
Pain threshold | 16 weeks
  Pain threshold will be measured at basline and 16 weeks and correlated to inflammatory markers and anisotropy

CONTACTS AND LOCATIONS:
Overall Officials: Smadar V Tourjman, MDCM, Principal Investigator — University of Montreal, Centre de recherche Fernand Seguin
Locations (1):
- Centre de Recherche Fernand-Seguin, Montreal, Quebec, Canada